CLINICAL TRIAL: NCT05346562
Title: Chronic Effects of Effective Oral Cannabidiol Delivery on 24-hour Ambulatory Blood Pressure and Vascular Outcomes in Treated and Untreated Hypertension: A Randomized, Placebo-controlled and Crossover Study
Brief Title: Oral Cannabidiol Effect on Blood Pressure in Hypertensive Patients
Acronym: HYPER-H21-4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Split, School of Medicine (Other)
Collaborators: Lexaria Bioscience Corp. (Industry); University of British Columbia (Other); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Zeljko Dujic, Professor, University of Split, School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2181-198-01-01-22-0002
Record Dates: First submitted 2022-04-06; First posted 2022-04-26 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Hypertension
Keywords: hypertension; cannabidiol; arterial stiffness
MeSH Terms: conditions — Hypertension | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cannabidiol, then Placebo (Experimental): Participant receive cannabidiol: 225 to 300 mg split over three times daily for the initial 2.5 weeks and 375 to 450 mg split over three times for the following 2.5 weeks. After two week washout, participant receives Placebo for five weeks (matching Cannabidiol tablets)
  Interventions: Dietary Supplement: Cannabidiol; Dietary Supplement: Placebo
- Placebo, then Cannabidiol (Experimental): Participant receive placebo tablets (matching Cannabidiol pills) for five weeks. After two week washout, Participant receive cannabidiol: 225 to 300 mg split over three times daily for the initial 2.5 weeks and 375 to 450 mg split over three times for the following 2.5 weeks.
  Interventions: Dietary Supplement: Cannabidiol; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cannabidiol — Cannabidiol tablets
Dietary Supplement: Placebo — Cannabidiol-matched placebo tablets

SUMMARY:
The objective of this randomized, placebo-controlled and crossover study is to extend the findings from the acute studies into more chronic administration of CBD in individuals with mild or moderate hypertension who are either untreated or receiving standard care therapy. The hypothesis is that the hypotensive effects of CBD will be apparent in both untreated and treated hypertension and reflected in improved vascular biomarkers and psychological well-being.

DETAILED DESCRIPTION:
Research Design A double-blind, placebo-controlled, cross-over pilot study in which 60 volunteers (aged 40-70 years) will visit to laboratory on six occasions following an overnight fast. All participants will provide written informed consent. Eligible participants will then be randomized. The sequence of conditions the participant will receive will be generated by a research randomizer web-service (https://www.randomizer.org) and participants will complete: 1) placebo-control and 2) DehydraTECHTM CBD (225 to 300 mg split over three times daily for the initial 2.5 weeks and 375 to 450 mg split over three times for the following 2.5 weeks) - see "dosing" below for further details . Following a two-week washout, volunteers will then repeat testing for another five weeks under the different condition. The study design, implementation and reporting will following the CONSORT guidelines, including the 25-item checklist and a flow diagram.

DehydraTECH is a patented formulation processing technology developed by Lexaria Bioscience Corp. that has been shown to enhance the performance of lipophilic beneficial compounds in oral ingestible products by way of increased rate and extent of intestinal bioabsorption and systemic uptake. DehydraTECH formulations have been prepared with a range of lipophilic molecules of interest and administered orally to animals and/or humans to investigate pharmacokinetic and pharmacodynamic performance attributes. For example, in young healthy humans, DehydraTECH technology has been studied in an oral CBD formulation and shown to result in higher and more rapid levels of delivery that was reflected in lower blood pressure when compared to positive controls with matching CBD concentrations (Patrician et al., 2019). Moreover, in volunteers with pre-hypertension, there were significant reductions in systolic, mean arterial blood pressure and arterial stiffness over an ambulatory 24-hr monitoring period following administration of oral DehydraTECH2.0 (150 mgs per 8 hours totalling 450 mgs) when compared to placebo. The DehydraTECH2.0 CBD was well tolerated with no ill-reported effects.

Both researchers and subjects will be blinded to the performed conditions on testing days by having a research associate who is not involved in any other aspect of the study supply the capsules according to the randomization schedule. When reporting to the laboratory in the morning will be in the fasted state (no food or drinks for at least 10 hours).

Visit 1 - Screening

On the initial visit potential participants will read through the information and consent form, ask any questions, and provide written informed consent. Following informed consent the participants will complete a customized Medical and Health Status Questionnaire that will be used to assess inclusion/exclusion criteria and prior history of medical conditions. Thereafter, the following questionnaires will be completed: Memory Assessment Clinic questionnaire(MAC-Q); Beck Anxiety Inventory (BAI); Perceived Stress Scale Questionnaire (PSS); Short Form 36 Health Survey Questionnaire (SF-36); Beck Depression Inventory (BDI); Global Physical Activity Questionnaire (GPAQ); State trait Anxiety Inventory (STAI); Big Life sodium calculator (BLSC). Sleep Questionnaires, including the Pittsburgh Sleep Quality Index (PSQI) and Epworth Sleepiness Scale (ESS); and the;); Stop-Bang Questionnaire (S-BANG).

Anthropometric and physiologic measurements will be collected (height, body weight, waist circumferences, bio-electrical impedance, blood pressure) for baseline participant characterization. After the completion of the screening procedures, the participants will be randomly assigned to one of the two experimental groups. Following randomization, participants will undergo first set of physiological, neuroimaging, sleep, and cognitive factors and will complete several lifestyle and psychological questionnaires. This battery of assessments will be completed again following either week 2.5 of week 5 before the washout period begins.

All subjects will be instructed to keep a food and physical-activity diary in the 24 h preceding the first laboratory visit and asked to replicate food consumption and physical activity as much as possible in the 24 h preceding subsequent visits. Subjects will be instructed to refrain from caffeine and alcohol-containing drinks for 6 and 12 h before each laboratory visit, respectively

Visit 2, 3 & 4 - Experimental Trials

The second visit will be scheduled at least 24 hours after the first visit to the laboratory and will require participants to be in the laboratory for <2 hours. Participants will report to the laboratory after an overnight fast (>10 hours) and around 07:30. Water intake will be measured and allowed ad-lib.

Dosing: For the initial 2.5 weeks, oral DehydraTECHTM CBD or the placebo control will be administered in the following doses during approx. 8-hr intervals for: a) males or females (who weigh>75 kg); 75mg at ~08:00, 75mg ~14:00 and 150mg ~22:00, total 300mg), b) males or females who weigh <75kg; (75mg at ~08:00, 75mg ~14:00 and 75mg ~22:00, total 225mg). For the final 2.5 weeks, upon confirmation of normal blood chemistry, the following doses during approx. 8-hr intervals for: a) males or females who weigh <100 kg; 75mg at ~8:00, 150 mg ~14:00 and 150mg ~22:00, total 375mg), b) males or females who weigh >100kg; (150 mg at ~8:00, 150 mg ~14:00 and 150mg ~22:00, total 450mg). The DehydraTECHTM CBD or the placebo control will be administered ~30 mins following consumption of a meal (to aid absorption). The timing of this dosing will be recorded by each subject and continue each day for the 5-week study duration. If a dose is missed, the subject will contact a member of the research team. he final daily dose (450 mg) will be the maximal dose approx. equally to 4.5 mg/kg/day. This dose is 2-4-fold less than the reported 1500mg/kg/day of CBD (or 10-20mg/kg/day) in the recent Phase 1 trial by Watkins and colleagues that revealed peak serum alanine aminotransferase values were above the upper limit of normal in 7 (44%) out of the 16 participants and exceeded international criteria for drug-induced liver injury in 5 (31%) of these participants (Watkins et al., 2021). The most common all-causality adverse events AEs by preferred term were gastrointestinal disorders, including diarrhea in eight (50%) participants and abdominal discomfort in five (31%) participants. Most of these AEs were first experienced during the CBD titration phase. AEs mild (31%) or moderate (50%) in severity.

Dosing diary and contingency for missed dosing: Each subject will be provided with a diary to confirm the timing of each daily dose of the CBD or placebo capsules. In the event of a missed dose, a maximum of one capsule (75mg) will be added to the next dose. The safety (lack of AEs) of acute dosing of 300 mg DehydraTECH2.0 CBD has been established; and previous studies have used much higher acute dosing without reports of related AEs (Sultan et al., 2020)

The 24-hour food log will be reviewed and a copy will be provided to subjects who will be asked to repeat the diet 24 hours before the following visit as closely as possible. Subjects will be reminded to not perform exercise or to consume alcohol 24 hours prior to the next visit. Subjects will return fasted to the laboratory approx. 17±2 days (~2.5 weeks) and 35±2 days (~5 weeks) after the second visit. Adherence to the 24-hour diet will be confirmed upon arrival in the laboratory and the snacks will be provided for each session. The subjects "dosing diary" will also be returned. Subjects will be instructed to identify any deviations in diet or dosing (from the food log and dairy) before beginning the previous trial.

Following the initial blood sample and questionnaires, subjects will then be instrumented with the 24-hour ambulatory blood pressure monitor (ABPM; TM-2430) that will be used to assess continuous blood pressure measurements away from the laboratory. The device will be set to take measurements every 30 minutes through the day (08:30-23:00) and every hour through the night (23:00-8:00). Subjects will be also instrumented with 24-hour ECG monitor. Subjects will also be asked to wear a Fitbit activity and sleep monitor (Fitbit Inc, San Francisco, CA, USA). This is a wrist-based device with a large organic light-emitting diode screen featuring heartrate monitoring and tracking of steps, distance, calories burned, floors climbed, active minutes, and sleep duration. The protocol will be the same as the other visit. Following the last visit and a 2-3 week washout period, subjects will receive one of the other two conditions.

Sample size Preliminary estimates of the effect sizes for improvement (lowering) of 24-hr ambulatory blood pressure following DehydraTECH2.0 are based on the results of the investigators' previous acute study that used similar active intervention and outcomes. This study will recruit a total of 70 participants, which will include a split of those who are either untreated or receiving standard care antihypertensive therapy. This power calculation, which is based on a sample size calculation formula for a mixed model for repeated measures data with attrition (Lu et al., 2008), provides 80% power to detect 0.4 standard deviation between-group difference for an average repeated measurement correlation of 0.6 and three repeated measurements, taking 20% attrition into consideration.

Statistical Analysis Continuous variables will be summarized with means ± standard deviation (SD) and/or 95% confidence intervals. Data will be analyzed for repeated measures analysis using either general or mixed linear models (with sex, body mass, medication and age as a co-variates). Significance will be set at 5% alpha and analyses will be calculated by SPSS version 21 software (IBM, Chicago, IL). A final analysis plan, which includes analyses of the secondary outcomes and strategies for handling missing/incomplete data, will be formalized by the biostatistician prior to breaking the blind. The data analysis will only begin once data collection is complete.

Significance The results of this study will help determine the effectiveness of Lexaria CBD technology as a novel anti-hypertensive agent, both in isolation and in combination with standard care therapy. Understanding new approaches to CBD delivery has major implications for more precise recommendations of CBD usage in health and disease states.

ELIGIBILITY:
Inclusion Criteria:

* Documented or measured elevated blood pressure (120/80 to 139/80 mmHg), mild (stage 1) hypertension (140/90 to 159/99 mmHg) or moderate (stage 2) hypertension (160/100 to 179/109 mmHg)
* Normal or overweight (body mass index 18.5 to 35.0 kg/m2)
* The female subjects are considered post-menopausal, and therefore not of reproductive potential, if they have not menstruated for at least 24 consecutive months in the absence of medications known to induce amenorrhea.
* Heterosexually active female subjects of reproductive potential must be on contraception management using at least one of the following methods while taking study drug and for 30 days following the last dose of study drug:

  * Barrier method of contraception [condoms (male or female), diaphragm, or cervical cap] with spermicide
  * IUD
  * Hormone-based oral, injectable, or implantable contraceptive
  * Bilateral tubal ligation/cauterization
  * Surgically sterile (hysterectomy or bilateral oophorectomy) or vasectomized male partner Undergo <150 minutes of moderate-to-vigorous activity per week Up to 40 subjects will be included who are not using anti-hypertensive therapy Up to 30 subjects will be included who are being treated with either (1) ACE inhibitors with or without diuretics or (2) ACE inhibitors with Calcium Channel blocker with or without diuretics.

Exclusion Criteria:

* Current smoker or using vapor-based products; or a medical or recreational cannabis user.
* Have kidney, liver disease (see below) or gastrointestinal disease (e.g., irritable bowel syndrome, celiac disease, Crohn's disease) or has had a cholecystectomy.
* Suffering from chronic diarrhea. (defined as >3 times loose / watery bowel movements per day lasting for more than 7 days; and occurring at least 4 times per year)
* Current diagnosis or history of any seizure disorder
* have diabetes
* cardiac instability / disease.
* are pregnant or breast feeding, or plan to become pregnant
* history of opioid use
* Dual blood pressure therapy other than ACE inhibitors with diuretic use and ACE inhibitors with Calcium Channel blocker with or without diuretics (e.g., ACE inhibitors with beta blockers)
* unwilling or unable to execute the informed consent documentation
* Liver disease, including, taking valproate, confirmed on baseline blood biochemistry - exclusion of subjects that have > 1.5 upper limit of normal (ULN) for ALT or AST, TBL >ULN at baseline determined by local reference population values in Croatia:

  * ULN for ALT 48 IU/L
  * ULN for AST 38 IU/L
  * ULN for ALP 142 IU/L
  * ULN for total bilirubin (TBL) 20 umol/L
  * ULN for GGT IU/L 55

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
24-hour ambulatory blood pressure | Through study completion, an average of 1 year
  Measured by ambulatory blood pressure monitoring system

SECONDARY OUTCOMES:
The burning of calories through physical activity | Through study completion, an average of 1 year
  Measured in kcal by wrist-based health & fitness tracker
Number of awakenings | Through study completion, an average of 1 year
  Measured by wrist-based health & fitness tracker
Total sleep time | Through study completion, an average of 1 year
  Measured by wrist-based health & fitness tracker
Total wake time | Through study completion, an average of 1 year
  Measured by wrist-based health & fitness tracker
Circulating cannabidiol | Through study completion, an average of 1 year
  Measured by venous blood sampling
Nitric oxide markers | Through study completion, an average of 1 year
  Measured by venous blood sampling
C-reactive protein concentration in serum | Through study completion, an average of 1 year
  Measured by venous blood sampling
Arterial stiffness | Through study completion, an average of 1 year
  Measured by pulse wave analysis
Volume of hippocampus | Through study completion, an average of 1 year
  Measured by MRI, T1-MPRAGE sequence
Blood flow through a. carotis interna | Through study completion, an average of 1 year
  Measured by MRI, 4D flow
Blood cholesterol concentration in serum | Through study completion, an average of 1 year
  Measured by venous blood sampling
Catestatin concentration in serum | Through study completion, an average of 1 year
  Measured by venous blood sampling
Liver enzymes in serum | Through study completion, an average of 1 year
  Measured by venous blood sampling
Heart rate | Through study completion, an average of 1 year
  Measured by 3-lead electrocardiogram
Salt intake | Through study completion, an average of 1 year
  Measured by Big life sodium calculator, range from 0 to 100 (higher score indicates higher salt intake)
Sleepiness | Through study completion, an average of 1 year
  Measured by Epworth sleepiness scale; range from 0 to 24 (higher score indicates higher sleepiness)
Geriatric depression | Through study completion, an average of 1 year
  Measured by Geriatric depression scale-short form; range from 0 to 15 (higher score indicates higher propensity for depression in geriatric population)
Physical activity | Through study completion, an average of 1 year
  Measured by Global Physical Activity Questionnaire; Total weekly MET-min is calculated in a following manner: (Minutes engaged in moderate-intensity activity each week X 4 MET) + (Minutes engaged in vigorous-intensity activity each week X 8 MET)
Memory | Through study completion, an average of 1 year
  Measured by Memory Complaint Questionnaire; range from 6 to 35 (higher scores indicate greater decline in memory)
Sleep quality | Through study completion, an average of 1 year
  Measured by Pittsburgh sleep quality index; range from 0 to 21 (higher score indicating worse sleep quality)
Perceived stress | Through study completion, an average of 1 year
  Measured by Perceived stress scale; range from 0 to 40 (higher score indicates higher perceived stress)
General health | Through study completion, an average of 1 year
  Measured by SF-36; range from 0 to 100 (higher scores indicate better health status)
Anxiety | Through study completion, an average of 1 year
  Measured by State-Trait Anxiety Inventory; range from 20 to 80 (higher scores indicates higher level of anxiety)
Obstructive sleep apnea risk | Through study completion, an average of 1 year
  Measured by STOP-BANG; range from 0 to 8 (higher scores indicate higher risk for OSA)
Depression | Through study completion, an average of 1 year
  Measured by Beck's Depression Inventory; range from 0 to 63 (higher score indicates higher level of depression)

CONTACTS AND LOCATIONS:
Overall Officials: Zeljko Dujic, MD, PhD, Principal Investigator — University of Split, School of Medicine
Locations (1):
- University of Split School of medicine, Split, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergamaschi MM, Queiroz RH, Chagas MH, de Oliveira DC, De Martinis BS, Kapczinski F, Quevedo J, Roesler R, Schroder N, Nardi AE, Martin-Santos R, Hallak JE, Zuardi AW, Crippa JA. Cannabidiol reduces the anxiety induced by simulated public speaking in treatment-naive social phobia patients. Neuropsychopharmacology. 2011 May;36(6):1219-26. doi: 10.1038/npp.2011.6. Epub 2011 Feb 9. PMID 21307846
- [Background] Granjeiro EM, Gomes FV, Guimaraes FS, Correa FM, Resstel LB. Effects of intracisternal administration of cannabidiol on the cardiovascular and behavioral responses to acute restraint stress. Pharmacol Biochem Behav. 2011 Oct;99(4):743-8. doi: 10.1016/j.pbb.2011.06.027. Epub 2011 Jul 12. PMID 21771609
- [Background] Jadoon KA, Tan GD, O'Sullivan SE. A single dose of cannabidiol reduces blood pressure in healthy volunteers in a randomized crossover study. JCI Insight. 2017 Jun 15;2(12):e93760. doi: 10.1172/jci.insight.93760. eCollection 2017 Jun 15. PMID 28614793
- [Background] Patrician A, Versic-Bratincevic M, Mijacika T, Banic I, Marendic M, Sutlovic D, Dujic Z, Ainslie PN. Examination of a New Delivery Approach for Oral Cannabidiol in Healthy Subjects: A Randomized, Double-Blinded, Placebo-Controlled Pharmacokinetics Study. Adv Ther. 2019 Nov;36(11):3196-3210. doi: 10.1007/s12325-019-01074-6. Epub 2019 Sep 12. PMID 31512143
- [Background] Sultan SR, Millar SA, England TJ, O'Sullivan SE. A Systematic Review and Meta-Analysis of the Haemodynamic Effects of Cannabidiol. Front Pharmacol. 2017 Feb 24;8:81. doi: 10.3389/fphar.2017.00081. eCollection 2017. PMID 28286481
- [Derived] Dujic G, Kumric M, Vrdoljak J, Dujic Z, Bozic J. Chronic Effects of Oral Cannabidiol Delivery on 24-h Ambulatory Blood Pressure in Patients with Hypertension (HYPER-H21-4): A Randomized, Placebo-Controlled, and Crossover Study. Cannabis Cannabinoid Res. 2024 Aug;9(4):979-989. doi: 10.1089/can.2022.0320. Epub 2023 Apr 21. PMID 37093160